CLINICAL TRIAL: NCT01247012
Title: A Randomized Controlled Trial of Minimization of Intralipid Versus Omegaven for the Treatment of Severe Cholestasis- A Pilot Trial
Brief Title: Minimization of IntraLipid Versus Omegaven
Acronym: MILOve
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Collaborators: Child and Family Research Institute (Other)
Responsible Party: Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MILOVE-134698
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Cholestasis; Parenteral Nutrition Associated Liver Disease (PNALD)
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipid minimization (Active Comparator)
  Interventions: Dietary Supplement: Lipid minimization
- Omegaven (Experimental)
  Interventions: Dietary Supplement: Omegaven

INTERVENTIONS:
Dietary Supplement: Omegaven — Omegaven 1g/kg/day until infant receiving full enteral feeds
  Arms: Omegaven
Dietary Supplement: Lipid minimization — 1g/kg/day daily until infant receiving full enteral feeds
  IF conjugated bili rises above 100, crossover to Omegaven (1gram/kg/day)
  Arms: Lipid minimization

SUMMARY:
Prolonged use of parenteral nutrition can lead to parenteral nutrition associated liver disease (PNALD). The purpose of this study is to determine the effect of treatment with a smaller amount lipid minimization) of our standard soybean oil based intravenous lipid emulsion (Intralipid) versus a fish-oil based lipid emulsion (Omegaven) in infants with severe cholestasis.

DETAILED DESCRIPTION:
Infants meeting eligibility will be randomized to receive either 1g/kg/day of Intralipid® 20% or 1g/kg/day Omegaven® 10%. Infants randomized to Intralipid® whose conjugated bilirubin level rises >100umol/L will be crossed over to receive 1g/kg/day Omegaven®. Monitoring includes liver function tests (AST, ALT,ALP, GGT, Conjugated Bilirubin), Fatty Acid Profile (RBC and serum fatty acids; triene/tetraene ratio), INR (coagulation profile) and cytokine measure (inflammatory markers).

ELIGIBILITY:
Inclusion Criteria:

* infants admitted to neonatal intensive care unit
* severe cholestasis, defined as conjugated bilirubin greater than 35
* receiving at least 60% calories by IV infusion and expected to require intravenous nutrition for at least an additional 28 days
* signed consent

Exclusion Criteria:

* hepatitis (TORCH or other viral infection)
* primary liver disease as etiology of cholestasis
* clinically severe bleeding not able to be managed with routine measures
* lethal congenital abnormalities
* congenital heart disease associated with right heart dysfunction

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | up to 1 year
  "Success" of the pilot trial will be determined by reaching the following criteria: 98.5% of subjects receive the modified lipid therapy within 12 to 24h of randomization; and/or 90% of subjects had their labs taken at the appropriate times as detailed by the study protocol.
Clinical endpoint | up to 1 year
  The proportion of subjects in each group that have a rise in conjugated bilirubin to or over 100 after randomization

SECONDARY OUTCOMES:
Total duration of parenteral nutrition | up to 1 year
Growth | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan Albersheim, MD, PhD, Principal Investigator — Children's & Women's Health Centre of BC; Avash J Singh, MD, Principal Investigator — Children's & Women's Health Centre of BC; Rebecca Sherlock, MD, Principal Investigator — Children's & Women's Health Centre of BC
Locations (1):
- Children's & Women's Health Centre of BC, Vancouver, British Columbia, Canada